CLINICAL TRIAL: NCT06028607
Title: A Study to Explore the Feasibility of Consumption of Specific Complex Amino Acid Supplementation in the Form of an Oral Gel With Additional Leucine (40%) and Vitamin D in Patients With Primary Ciliary Dyskinesia: a Feasibility Study
Brief Title: Feasibility of Consumption of Nutritional Supplementation in Primary Ciliary Dyskinesia
Acronym: (PCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Professor Daniel G Peckham, Professor of Respiratory Medicine, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Version 1.0
Record Dates: First submitted 2023-08-24; First posted 2023-09-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Intervention Model Description: All service users will be approached for inclusion in feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population (Other): Participants will be recruited and consented as part of routine care. All will trial supplement initially and have standard and additional measures taken. they will be followed up at month 1 and 2 collecting the primary outcomes (acceptability/palatability and dietary intake) and all initial measures repeated at month 3.
  Each participant will receive 3 months supply of gels to consume 2 per day.
  Interventions: Dietary Supplement: QD-27

INTERVENTIONS:
Dietary Supplement: QD-27 — Oral Protein gel with greater Leucine proportion and vitamin D Consumption of 2 each day for 3 months to be taken at breakfast and lunch

SUMMARY:
Feasibility study to understand and gain preliminary information on tolerability and palatability of an oral nutritional supplement gel in a clinical Primary Ciliary Dyskinesia population. To determine if dietary intake is affected by the consumption of the nutritional supplement.

Explore possible future outcome measures that could be important in determining impact of this nutritional intervention on this patient group.

Participants will be provided with the gel supplements and alongside will have other standard and non standard care measures assessed lung function (FEV1%) number of exacerbation's during study period vitamin D status Bio impedance analysis (BIA) skin-fold measures (e.g. Tricep Skin-fold (TSF) Mid upper arm circumference (MUAC) Handgrip strength (HGS) quality of life measures 6-minute walking tests. Hypothesis Patients with PCD can successfully consume 2 gel supplements per day for a period of 3 months with no effect on dietary intake.

DETAILED DESCRIPTION:
This is a single site study taking place in a regional PCD clinic. Participants are screened via patient online data system by lead consultants and contacted via telephone to outline study and provide information and contact for queries. participant information sheet and pre-test guidance to be sent to participant prior to next scheduled clinic appointment.

Participants attend their usual clinic appointments where routine care measures are completed by healthcare assistants and lead consultants. They then have opportunity to ask study coordinator any questions and complete consent for additional measures to be recorded.

This is followed by a trial of the supplement to check for immediate tolerance followed by completion of consent to partake in study and initial palatability and acceptability records.

3 month supply of supplement is provided along with storage and consumption instructions (consume 1 at breakfast and 1 at lunch) a waste box to retain consumed sachets and record time of consumption. Additional telephone appointment made for 1 month to collect further palatability and acceptability along with dietary 24 hour recall.

Participant is contacted via telephone at month 1 and 2 to recheck tolerability, acceptability, palatability and dietary intake. Participant can withdraw at any time if unable to continue to tolerate gel supplement.

Participant returns to clinic at month 3 to repeat all standard measures, additional outcomes and palatability, acceptability and dietary intake.

participant has completed study offered further dietary support through usual clinic route with registered dietitian.

Participants can withdraw from the study at any point without giving any reason. Any data collected from them up until that point can be used in analysis.

As this is a feasibility study a sample size calculation is not required. The PCD population within the regional clinic at time of recruitment is 54. All patients with PCD will be approached for inclusion in this feasibility if they meet the inclusion criteria until minimum number of 15 and maximum of 20 is reached.

ELIGIBILITY:
Inclusion Criteria:

* People aged 17 or over with a confirmed diagnosis of Primary ciliary dyskinesia PCD (nasal brushings)
* People who attend the Leeds Regional PCD Clinics
* People who have capacity to give informed consent

Exclusion Criteria:

* People who are pregnant
* Those with existing co-morbidities such as malignancy
* People with connective tissue disorders and immunoglobulin deficiencies
* People with renal insufficiency r

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage consumption of supplement gels | 3 months
  To measure through percentage (%) consumed by return of empty sachets over period of three months for each participant
Assessment of palatability of supplement gels | 3 months
  To measure using hedonic rating scale (like a lot, like a little, neither like nor dislike, dislike a little, dislike a lot) the appearance, aroma, taste, sweetness, texture mouth feel over the study period of 3 months for each participant
Measurement of dietary intake | 3 months
  To collect dietary intake at monthly intervals (baseline, one, two and three) using multiple pass 24 hour recalls conducted through face to face and telephone interviews at each time point recording all food and drink consumption. This is then analysed via Nutritics software, for each participant

SECONDARY OUTCOMES:
Lung Function (Forced Expiratory Volume1 %, Forced Vital Capacity %) | 3 months
  Determine if any changes occur during 3-month period of supplementation
Body Mass Index | 3 months
  Weight and height will be combined to report BMI in kg/m2
Medical Research Council (MRC) breathlessness score | 3 months
  Will be assessed at initial and end points using the degree of breathlessness related activity. Scale is 1-5 (not troubled by breathless except on strenuous exercise to too breathless to leave the house or breathless when dressing and undressing) therefore the higher the score the worse the outcome
Vitamin D levels | 3 months
  To determine any changes during supplementation period
Number of infections over study period | 3 months
  Recorded as part of routine care the number of infections requiring antibiotic treatment either intravenous or oral) over the study period
Quality of life outcome SF-36 questionnaire | 3 months
  Completion of SF-36 quality of life questionnaire questionnaire which is used to determine generic health concepts of functional status and wellbeing. Completed at baseline and end of study period. The higher the score the better the health outcomes
Quality of Life outcome St Georges Respiratory Questionnaire | 3 months
  Completion of St Georges Respiratory questionnaire designed to measure health impairment in respiratory conditions. The results are calculated out of 100 with 100 being the worst possible outcomes and 0 the best.
Habitual activity estimation scale (HAES) | 3 months
  HAES scale which establishes daily activity levels at baseline and end of study for one typical weekday and one typical weekend day and using percentage of time spent on those activities out of 100%.
Hand grip strength dynamometry | 3 months
  Measurement of muscle functionality using hand grip dynamometer recorded as kg/f (kilograms of force)
Tricep skinfold measure | 3 months
  To determine any changes during supplementation period. Measured in millimetres using Harpenden skinfold calipers
Mid upper arm circumference | 3 months
  To determine any changes during supplementation period measured in centimetres, measured using an identified mid point between the acromion and olecranon processes using a tape measure
Six minute walk tests | 3 months
  To determine any changes during supplementation period
Bio electrical impedance analysis | 3 months
  Measure the electrical resistance of tissue to determine skeletal muscle mass reported as percentages and kilograms of participants at baseline and end point
Bio electrical impedance analysis | 3 months
  Measure the electrical resistance of tissue to determine fat mass (FM), reported as percentages and kilograms of participants at baseline and end point
Bio electrical impedance analysis | 3 months
  Measure the electrical resistance of tissue to determine fat free mass (FFM) reported as percentages and kilograms of participants at baseline and end point

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Peckham, Principal Investigator — Univeristy Of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018